CLINICAL TRIAL: NCT00285363
Title: Quality of Life Among Children and Adolescents With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Unable to reconcile record due to age
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 04 05-052E; CMCC grant
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: cancer; quality of life; adolescents
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This descriptive study aims to allow children and adolescents who have cancer to self-evaluate their quality of life. It is hypothesized that treatment affects quality of life in the areas of physical and social functioning. It is further hypothesized that these effects dissipate within 6 months after treatment is completed.

DETAILED DESCRIPTION:
Study participants will include all children and adolescents (aged 7 to 21 years old) currently receiving care from the Hematology/Oncology Clinic at the CMHC, which will serve as the study site. These individuals will be identified by the health care professionals working in the clinic. Specific study criteria will include only those individuals who (1) can read or write in the English language (due to limited availability of translators); (2) appear to not possibly suffer psychological harm by participating (as determined by any health care professional working in the Clinic); and (3) do not have a health condition and/or medical need that supersedes study participation. The weekly list of appointments will be reviewed by the researchers who already work in the Clinic for appropriateness (JH, JB and KS). To prevent participation coercion, solicitation for participation will be provided through the Child Life Specialist (CLS). The CLS is known to each participant and will function as a data collector for this study.

ELIGIBILITY:
Inclusion Criteria:Study participants will include all children and adolescents (aged 7 to 21 years old) currently receiving care from the Hematology/Oncology Clinic at the CMHC, which will serve as the study site. These individuals will be identified by the health care professionals working in the clinic. Specific study criteria will include only those individuals who (1) can read or write in the English language (due to limited availability of translators); (2) appear to not possibly suffer psychological harm by participating (as determined by any health care professional working in the Clinic); and (3) do not have a health condition and/or medical need that supersedes study participation. -

Exclusion Criteria: (1) Those electing not to participate; (2) those with no guardian available to consent or (3) those not yet diagnosed with a cancer condition.

-

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Ward-Smith, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States